CLINICAL TRIAL: NCT04648709
Title: Evaluation and Longitudinal Follow-up of Biomarkers Predictive of Severe Forms of COVID-19
Acronym: COVIMMUNITY
Status: Terminated | Type: Observational
Why Stopped: The development and generalisation of vaccination led to a significant drop in the number of patients meeting the inclusion criteria.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH207; 2020-A02943-36 (Other: ANSM)
Record Dates: First submitted 2020-11-27; First posted 2020-12-01 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-02

CONDITIONS: Covid19
Keywords: T cells; B cells; immune response; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Enzyme-Linked Immunospot Assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- asymptomatic patients: asymptomatic patients with PCR-positive PCR
  Interventions: Diagnostic Test: ELISPOT; Diagnostic Test: QUANTIFERON
- mild symptoms patients: patients with mild symptoms and PCR positive
  Interventions: Diagnostic Test: ELISPOT; Diagnostic Test: QUANTIFERON
- seriously symptomatic patients: seriously symptomatic patients with PCR positive
  Interventions: Diagnostic Test: ELISPOT; Diagnostic Test: QUANTIFERON
- patients in resuscitation: patients in resuscitation with positive PCR
  Interventions: Diagnostic Test: ELISPOT; Diagnostic Test: QUANTIFERON
- heathly volunteer: heathly volunteer as control
  Interventions: Diagnostic Test: ELISPOT; Diagnostic Test: QUANTIFERON

INTERVENTIONS:
Diagnostic Test: ELISPOT — measure of immune response by ELISPOT
Diagnostic Test: QUANTIFERON — measure of immune response by QUANTIFERON

SUMMARY:
Current data in the literature demonstrate that the immune response to CoV-2-SARS is much more complex than initially assumed. In fact, beyond the humoral response, including the existence of neutralizing CAs, the adaptive lymphocyte T-type immune response also appears to play an important role in controlling the infection and reducing the severity of the disease. At this stage, the analysis of this T response is still rudimentary and underdeveloped, but it seems crucial to be able to analyze it effectively in COVID-19 patients, which could help predict the evolution of the infection. It is also currently difficult to know the evolution of this response over time and especially after the resolution of the infection.

To this end, we will analyze the T lymphocyte response (ELISPOT and QUANTIFERON) based on the secretion of IFN (Th1) and IL-4 (Th2) by CoV-2-SARS specific T cells from COVID-19 patients. We will compare the T response to the quality of the systemic and mucosal humoral response. Finally, we will evaluate in parallel two new biomarkers of the severity of COVID-19: plasma calprotectin and the presence of antibodies to type 1 IFN antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Social security affiliation
* Signed informed consent
* Patients with COVID infection documented by PCR and/or antigenic testing
* Patients belonging to the following groups:

  * asymptomatic patients with PCR-positive PCR
  * patients with mild symptoms and PCR positive
  * seriously symptomatic patients with PCR positive
  * patients in resuscitation with positive PCR
  * Healthy individuals as controls

Exclusion Criteria:

* haemoglobin < 8g/dL
* Pregnancy, breastfeeding woman
* Patient vaccinated within 15 days prior to inclusion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with COVID infection documented by PCR and/or antigenic testing will be included.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
T cell immune response | from baseline to 18 months
  Characterize T-cell immune response in patient with COVID 19 infection

SECONDARY OUTCOMES:
B cell immune response | from baseline to 18 months
  Characterize B-cell immune response in patient with COVID 19 infection
Platelet immune response | from baseline to 18 months
  Characterize platelet immune response in patient with COVID 19 infection
Immune response and chronic forms | from baseline to 18 months
  Determine if there is a correlation between the pattern of immune response and the risk of reinfection or with persistence of symptoms in chronic forms of COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Paul, PHD, Study Director — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No